CLINICAL TRIAL: NCT03985150
Title: Biomechanical Characterization of Atherosclerotic Arterial Tissue of the Femoralis Superficialis
Brief Title: Biomechanical Analysis of Arterial Tissue From Patient Suffering From Peripheral Artery Disease in the Lower Limb
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S62776
Record Dates: First submitted 2019-05-27; First posted 2019-06-13 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The superficial femoral artery will be collected from the amputated limb
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomechanical analysis of femoralis superficialis atherosclerotic tissue — Tissue collection during above-knee amputation; mechanical testing of tissue; microstructural testing of tissue
Radiation: CT or MR angiogram — Obtaining in vivo geometry of diseased artery

SUMMARY:
The current treatment approaches for peripheral artery disease are largely unsatisfactory. Therefore, diseased tissue will be collected as well as patient-specific arterial geometries. The tissue will be tested microstructurally and mechanically to obtain data required to optimize treatment methods through in silico modeling.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a severe cause of morbidity in patients. Common treatment approaches are too often still unsatisfactory. Angioplasty is commonly followed by restenosis, caused by overloading of the arterial tissue. This study is aimed at improving this treatment approach through the in silico simulation of arterial remodeling after balloon expansion. Such simulations require the input of a patient-specific geometry and the mechanical properties of (diseased) arterial tissue.

Patients scheduled for an above knee lower limb amputation due to critical ischemia will be recruited in this study. After the surgery, the femoralis superficialis will be collected, as well as the CT or MR angiogram obtained before the surgery. The arterial tissue will be mechanically tested to obtain material properties and the medical image will be used to determine the arterial geometry. A correlation study will be carried out to explore the possibility of including a predictive simulation of the restenosis outcome of balloon angioplasty in the clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from critical ischemia in the lower limb and undergoing above-knee amputation

Exclusion Criteria:

* The presence of any feature that will prevent tissue collection after the amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from peripheral arterial disease
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Biaxial stress-stretch curves of diseased superficial femoral arterial tissue from planar biaxial tension tests. | up to 3 years
  Planar biaxial tension tests will be performed on the collected tissue. The results of these tests, in the form of stress-stretch curves, will be fitted to existing or to be developed constitutive models describing the mechanical behavior of arterial tissue.
Axial force and diameter curves in function of pressure from extension-inflation tests on diseased superficial femoral arterial tissue. | up to 3 years
  Extension-inflation tests will be performed on the collected tissue. The results of these tests, in the form of axial force and diameter curves, will be fitted to existing or to be developed constitutive models describing the mechanical behavior of arterial tissue.
Reaction force curves in function of indentation depth from indentation tests on diseased superficial femoral arterial tissue. | up to 3 years
  Indentation tests will be performed on the collected tissue. The results of these tests, in the form of reaction force versus indentation depth curves, will be fitted to existing or to be developed constitutive models describing the mechanical behavior of arterial tissue.

SECONDARY OUTCOMES:
Microstructural composition of diseased superficial femoral arterial tissue from histological analyses | up to 3 years
  Histological images will be analyzed to obtain the microstructural organization and composition of the collected tissue samples.
Microstructural composition of diseased superficial femoral arterial tissue from microCT analyses | up to 3 years
  MicroCT images will be analyzed to obtain the microstructural organization and composition of the collected tissue samples.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven campus Gasthuisberg, Leuven, Belgium